CLINICAL TRIAL: NCT00952003
Title: Phase II Study of Oxaliplatin / Irinotecan / Bevacizumab Followed by Docetaxel / Bevacizumab in Inoperable Locally Advanced or Metastatic Gastric Cancer Patients
Brief Title: Oxaliplatin/Irinotecan/Bevacizumab Followed by Docetaxel/Bevacizumab in Inoperable Locally Advanced or Metastatic Gastric Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Pfizer (Industry); Sanofi (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT GASTRIC-3
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Gastric Cancer; Unresectable
Keywords: Avastin; Campto; Oxaliplatin; Taxotere
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Irinotecan; Bevacizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- interventional arm (Experimental): Oxaliplatin, Irinotecan and Bevacizumab for 3 cycles followed by Docetaxel and Bevacizumab for a further 3 cycles. Upon completion of the combination therapy cycles Bevacizumab will be continued until progression.
  Interventions: Drug: Oxaliplatin, Irinotecan, Bevacizumab, Docetaxel

INTERVENTIONS:
Drug: Oxaliplatin, Irinotecan, Bevacizumab, Docetaxel

SUMMARY:
The primary objective of this study is to determine the efficacy of an Oxaliplatin / Irinotecan / Bevacizumab therapy followed by Docetaxel / Bevacizumab therapy followed by Bevacizumab until progression in the treatment of locally advanced metastatic gastric cancer, in terms of response rates (complete or partial response, determined by radiologic evaluation according to Response Evaluation Criteria in Solid Tumors (RECIST)).

Secondary objectives Secondary Objective: To determine the safety profile of a an Oxaliplatin/Irinotecan/Bevacizumab therapy followed by Docetaxel/Bevacizumab therapy followed by Bevacizumab until progression in terms of qualitative and quantitative toxicities from first study treatment dose until completion of study treatment due to progression or for any other reason.

Secondary Objective: To evaluate the study population with respect to the following: overall survival (from treatment start until death from any cause) and progression free survival (from treatment start until progression or death from any cause).

DETAILED DESCRIPTION:
This is a non-randomized, multicenter, open-label, single-arm Phase II study in patients with inoperable histologically proven inoperable locally advanced or metastatic gastric cancer. Eligible patients must be therapy naïve and have received no previous chemotherapy or immune therapy for their inoperable gastric cancer. Neo/Adjuvant Chemotherapy or adjuvant Chemo/Radiotherapy are allowed. A total of 40 evaluable patients will be recruited and evaluated for efficacy and safety of a sequential chemoimmunotherapy combination regime.

Overall Study Design:

Eligible patients will receive Oxaliplatin, Irinotecan and Bevacizumab for 3 cycles followed by Docetaxel and Bevacizumab for a further 3 cycles. Upon completion of the combination therapy cycles Bevacizumab will be continued until progression. Safety assessments will be conducted in 4-weekly intervals; efficacy assessments will be conducted at 12 weekly intervals, at completion of every third treatment cycle.

This study is expected to start in Q1 2009. The last patient is expected to enter the study in Q2 2010, following an 18 month recruitment period. Taking into account treatment duration the study is expected to end in Q4 2010. Study end will be at Last Subject Last Visit at Final Staging upon disease progression. Follow-up after Last Subject Last Visit will be conducted according to local standard of care thereafter, and is not part of study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histologically proven gastric adenocarcinoma
* Measurable or evaluable, inoperable locally advanced or metastatic disease. Presence of at least one measurable lesion according to RECIST criteria.
* No previous palliative chemotherapy and/or immunotherapy
* Life expectancy of more than 3 months
* Age ≥ 18 years.
* ECOG performance status 0 - 2
* Ability to understand and comply with requirements of study protocol and trial participation
* Patients of either sex are eligible for study entry. Women of childbearing potential must have a negative pregnancy test at screening and must use effective contraception (e.g. intrauterine device (IUD), birth control pills, or barrier device) beginning 2 weeks prior to first dose of study drug until 6 months after the final dose of study drug.
* Hematological status:

Leucocytes ≥ 3 x 109/l Platelets ≥ 100 x 109/l •Renal function: Serum creatinine: ≤ 1.5 x upper normal limit of normal (ULN)

•Hepatic function: AST and ALT: < 2.5 x ULN or < 5 x ULN if hepatic metastases are present Alkaline phosphatase: < 2.5 x ULN or < 5 x ULN if hepatic metastases are present Total bilirubin level ≤ 1.5 x ULN

* Patient must have an INR ≤ 1.5 and aPTT ≤ 1.5 x ULN within 7 days prior to randomisation
* Baseline evaluations performed before treatment start: clinical and blood evaluations no more than 7 days prior to planned first course; tumoral assessment (CT scan or MRI) no more than 4 weeks prior to planned first course

Exclusion Criteria:

* Pregnant or lactating women.
* Women of child-bearing potential and men not using effective contraception.
* Concurrent cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy) or
* Neo/Adjuvant treatment with Irinotecan and/or docetaxel and/or Bevacizumab
* Patients with locally advanced disease who are candidates for curative therapy (including operation and/or chemotherapy and/or radiotherapy).
* Prior history of chronic enteropathy, chronic diarrhea, unresolved bowel obstruction/ subobstruction, or extensive abdominopelvic radiation therapy.
* Previous malignancy other than gastric cancer in the last 5 years except curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix.
* Evidence of CNS metastasis at baseline. A CT or MRI scan within 28 days prior to randomisation is mandatory to exclude CNS involvement in case of clinical suspicion of CNS metastasis.
* Peripheral neuropathy (NCI CTC grade ≥ 1).
* Inadequate renal function:
* adequate renal function:ould be ≥ 60 mL/min. The Cockroft and Gault formula is recommended for calculation of creatinine clearance. Patients with a creatinine clearance just below 60 ml/min may be eligible if a measured creatinine clearance (based on 24 hour urine collection or other reliable method) is ≥ 60 mL/min.
* Urine dipstick for proteinuria should be < 2+. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hour urine collection and must demonstrate < 1 g of protein/24 hr.
* Serious medical or psychiatric disorders that would interfere with the patient's informed consent or compliance with the requirements of the protocol or that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.
* Active bacterial, viral or fungal infection (including acute or chronic-active infection with HBV or HCV).
* Acute intra abdominal inflammatory process.
* Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) or clinically significant (i.e. active) cardiovascular disease, for example cerebrovascular accidents (≤ 6 months prior to randomisation), myocardial infarction (≤ 6 months prior to randomisation), unstable angina, New York Heart Association Grade II or greater congestive heart failure, or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment.
* Prior history of hypertensive crisis or hypertensive encephalopathy.
* Evidence of tumour invading major blood vessels on imaging. The investigator or the local radiologist must exclude evidence of tumour that is fully contiguous with, surrounding, or extending into the lumen of a major blood vessel (e.g. pulmonary artery or superior vena cava).
* Serious uncontrolled coagulation disorder or thrombo-embolic complications (history of embolisms or thromboses) within 6 months prior to study start or history of inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* Major surgical procedures within 4 weeks prior to study entry or planned major surgical procedures throughout the course of the study. Patients must have fully recovered from any surgical procedures conducted prior to 4 weeks before study entry.
* Minor surgery, including insertion of an indwelling catheter, within 48 hours prior to the first bevacizumab infusion.
* Concurrent or recent (within 10 days) anticoagulant therapy. Prophylactic use of anticoagulants is allowed.
* Chronic daily treatment with aspirin (> 325 mg/day) or clopidogrel (> 75 mg/day).
* Chronic daily treatment with oral corticosteroids (dose of > 10 mg/day methylprednisolone equivalent). Inhaled steroids and short courses of oral steroids for anti-emesis or as an appetite stimulant are allowed.
* Known history of Deep Vein Thrombosis (DVT) and/ or pulmonary embolism (PE).
* Non-healing wound, active peptic ulcer or bone fracture.
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrolment or active gastrointestinal bleeding.
* Concurrent treatment with an investigational drug or participation in another clinical trial.
* Contraindications for the study regimen or known hypersensitivity to the study drugs or to Chinese hamster ovary cell products or to other recombinant human or humanised antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2014-10-22 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
To determine efficacy in terms of response rate according to RECIST criteria | 3-6 months

SECONDARY OUTCOMES:
Safety of treatment | 3-6 months
To determine median progression-free survival times following treatment with a chemoimmune therapy | 3 - 6 months
To determine overall survival time following treatment with a chemoimmune therapy | 3 - 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, Prof.Dr., Study Chair — AGMT Arbeitsgemeinschaft Medikamentöse Tumortherpie gemeinnützige GmbH
Locations (7):
- Austria (7):
  - Universitätsklinik Innsbruck, Innsbruck
  - A.ö. Landeskrankenhaus Leoben, Leoben
  - Krankenhaus der Stadt Linz, Linz
  - Universitaetsklinik f. Innere Medizin III, Salzburg
  - Universitätsklinik Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
  - BKH Zams, Zams